CLINICAL TRIAL: NCT04930809
Title: Open-label Study to Evaluate the Pharmacokinetics and Safety of VER-01after Single and Multiple Administration of Different Doses to Healthy Volunteers
Brief Title: Single and Multiple Dose Study of VER-01 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertanical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VER-PK-001
Record Dates: First submitted 2021-05-24; First posted 2021-06-18 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: THC; Tetrahydrocannabinol; Cannabis; Pharmacokinetics
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- VER-01 single dose (2.5 mg THC) (Experimental): PK profile is investigated after oral intake of a single dose VER-01 corresponding to 2.5 mg THC (Group A).
  Interventions: Drug: VER-01
- VER-01 single dose (5 mg THC) (Experimental): PK profile is investigated after oral intake of a single dose VER-01 corresponding to 5 mg THC (Group B).
  Interventions: Drug: VER-01
- VER-01 single dose (10 mg THC) (Experimental): PK profile is investigated after oral intake of a single dose VER-01 corresponding to 10 mg THC (Group C).
  Interventions: Drug: VER-01
- VER-01 single dose (20 mg THC) (Experimental): PK profile is investigated after oral intake of a single dose VER-01 corresponding to 20 mg THC (Group D).
  Interventions: Drug: VER-01
- VER-01 multiple dose (5 mg THC) (Experimental): PK profile is investigated after oral intake of VER-01 corresponding to 5 mg THC in the morning and 5 mg THC in the evening on 4 consecutive days (Group E).
  Interventions: Drug: VER-01
- VER-01 multiple dose (10 mg THC) (Experimental): PK profile is investigated after oral intake of VER-01 corresponding to 10 mg THC in the morning and 10 mg THC in the evening on 4 consecutive days (Group F).
  Interventions: Drug: VER-01
- VER-01 multiple dose (12.5 / 20 mg THC) (Experimental): PK profile is investigated after oral intake of VER-01 corresponding to 12.5 mg THC in the morning and 20.5 mg THC in the evening on 4 consecutive days (Group F).
  Interventions: Drug: VER-01

INTERVENTIONS:
Drug: VER-01 — standardised cannabis extract (containing 21 mg THC per gram drug product)

SUMMARY:
Evaluation of pharmacokinetics, tolerability and safety of VER-01 in healthy volunteers

DETAILED DESCRIPTION:
Determination of the single and multiple dose pharmacokinetic profile of VER-01 in healthy volunteers.

Single dose: 6 subjects each will receive VER-01 corresponding to 2.5 mg (Group A), 5 mg (Group B), 10 mg (Group C) or 20 mg THC (Group D) in the morning.

Multiple dose: 6 Subjects each receive VER-01 corresponding to 5 mg (Group E) or 10 mg (Group F) THC in the morning and in the evening on 4 consecutive days. A third group (Group G) receives VER-01 corresponding to 12.5 mg THC in the morning and 20 mg THC in the evening on 4 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers
* Age: 18-45 years
* BMI: 19-30 kg/m²
* Body weight ≥ 50 kg
* volunteers in good general condition based on medical history, physical examination, resting ECG and clinical laboratory tests
* Willingness of men to use a reliable method of contraception and not to donate sperm during and at least 3 months after the last intake of the study product
* Understanding of the German language, ability to give consent and compliance
* The subject has understood the instructions to avoid changes in lifestyle and eating habits
* Signed patient information and written informed consent form of the study participant

Exclusion Criteria:

* Consumption of cannabis-based products within 30 days prior to study start
* Well-known strong adverse events in connection with cannabis consumption
* Known allergy to cannabis, sesame seeds, or derivative products
* alcohol/drug/medication abuse or physical dependence on opioids, barbiturates, amphetamines, cocaine or benzodiazepines within the last 10 years or current intake of methadone
* Positive drug test for illegal substances and/or alcohol test at time T0
* Heavy smokers (>10 cigarettes/day)
* Heavy caffeine consumers (>450 mg caffeine/day equal to approx. 5-6 cups of filter coffee)
* Drastic change in diet within 30 days before study start
* Mental illness (psychoses, schizophrenia, bipolar disorder, severe depression, anxiety disorder, suicide)
* Mental illness (psychoses, schizophrenia, bipolar disorder, severe depression, anxiety disorder, suicide) in a first-degree relative (parents and children)
* subjects with orthostatic hypotension during screening (drop in systolic blood pressure by ≥20 mmHg after change of position)
* Cardiovascular event within the last 3 months, untreated hypertension, untreated hypothyroidism, surgery within the last 2 months
* cardiac insufficiency
* Subjects with a serious disease or disorder which, in the opinion of the investigator, does not allow safe participation in the study from a medical point of view
* Intake of prescription drugs within the last 14 days, over-the-counter test products within the last 7 days before the start of the study or during the study period
* Eating of grapefruit products is not allowed during the study and 10 days before the first intake of the study product
* Participation in another clinical trial in the period of 90 days before the start of the trial
* Existing desire to have children or planned sperm donation (within the duration of the study and 3 months after end of the study)
* Planned blood donation
* No ability to consent
* Subject is in a dependency/employment relationship with the sponsor or investigator or other persons who may be under pressure.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC] - AUC 0-t | Group A-D: Day 1; Group E-G: Day 1 and 4
  Analysis of the AUC 0-t (AUC from time 0 to 24 hours) of THC over a defined period of time.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC] - AUC 0-∞ | Group A-D: Day 1; Group E-G: Day 1 and 4
  Analysis of AUC 0-∞ (AUC from time 0 extrapolated to infinity) of THC over a defined period of time.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC] - C max | Group A-D: Day 1; Group E-G: Day 1 and 4
  Analysis of C max (maximum plasma concentration) of THC over a defined period of time.

SECONDARY OUTCOMES:
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - AUC 0-t | Group A-D: Day 1; Group E-G: Day 1 and 4
  Analysis of AUC 0-t (AUC from time 0 to 24 hours) of 11-OH-THC and THC-COOH over a defined period of time.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - AUC 0-∞ | Group A-D: Day 1; Group E-G: Day 1 and 4
  Analysis of AUC 0-∞ (AUC from time 0 extrapolated to infinity) of 11-OH-THC and THC-COOH over a defined period of time.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - C max | Group A-D: Day 1; Group E-G: Day 1 and 4
  Analysis of C max (maximum plasma concentration) of 11-OH-THC and THC-COOH over a defined period of time.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - λ z | Group A-D: Day 1; Group E-G: Day 1 and 4
  Analysis of λ z (terminal elimination constant) of THC, 11-OH-THC and THC-COOH over a defined period of time.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - t 1/2 | Group A-D: Day 1; Group E-G: Day 1 and 4
  Analysis of t 1/2 (elimination half-life) of THC, 11-OH-THC and THC-COOH over a defined period of time.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - T max | Group A-D: Day 1; Group E-G: Day 1 and 4
  Analysis of T max (time to reach Cmax) of THC, 11-OH-THC and THC-COOH over a defined period of time.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - C L/F | Group A-D: Day 1; Group E-G: Day 1 and 4
  Analysis of C L/F (plasma clearance) the pharmacokinetic profile of THC, 11-OH-THC and THC-COOH over a defined period of time.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - V area/F | Group A-D: Day 1; Group E-G: Day 1 and 4
  Analysis of V area/F (volume of distribution) of THC, 11-OH-THC and THC-COOH over a defined period of time.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, Professor, Principal Investigator — University of Medicine in Vienna - Department of Clinical Pharmacology
Locations (1):
- University of Medicine in Vienna - Department of Clinical Pharmacology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No